CLINICAL TRIAL: NCT05711576
Title: The Effect of Non-surgical Mechanical Debridement With or Without Full-mouth Disinfection in the Treatment of Peri-implant Mucositis. A Randomized Placebo-controlled Clinical Trial
Brief Title: Non-surgical Mechanical Debridement With or Without Full-mouth Disinfection in the Treatment of Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Principal Investigator, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 150/2679/2022/PO
Record Dates: First submitted 2022-12-26; First posted 2023-02-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Intervention Model Description: At baseline, 1, 3, 6 months, full-mouth plaque score (FMPS), full-mouth bleeding score (FMBS), probing depth (PD), bleeding on probing (BOP), modified gingival index (mGI), and modified plaque index (mPlI) were assessed.
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-surgical sub-marginal peri-implant instrumentation (NSPI) with placebo mouthwash (Placebo Comparator): Patients received a one-session of non-surgical sub-marginal peri-implant instrumentation (NSPI) with placebo mouthwash
  Interventions: Other: Placebo mouthwash
- non-surgical sub-marginal peri-implant instrumentation (NSPI) with FMD (Active Comparator): Patients received a one-session of non-surgical sub-marginal peri-implant instrumentation (NSPI) with full-mouth disinfection approach (FMD).
  Interventions: Other: Full mouth disinfection

INTERVENTIONS:
Other: Placebo mouthwash — Patients were treated with non surgical peri-implant mucositis therapy with non-surgical sub-marginal peri-implant instrumentation plus the use of a placebo mouthwash
  Arms: non-surgical sub-marginal peri-implant instrumentation (NSPI) with placebo mouthwash
Other: Full mouth disinfection — Patients were treated with non surgical peri-implant mucositis therapy with non-surgical sub-marginal peri-implant instrumentation plus the use of full mouth disinfection (FMD) approach
  Arms: non-surgical sub-marginal peri-implant instrumentation (NSPI) with FMD

SUMMARY:
To evaluate the naturally occurring peri-implant mucositis (PM) treatment by means of non-surgical sub-marginal peri-implant instrumentation (NSPI) with or without full-mouth disinfection approach (FMD). Specifically, the primary outcome of the present study compared the efficacy of NSPI and full-mouth disinfection (FMD) with respect to NSPI and placebo in the treatment of PM at 6 months follow-up. The secondary outcome evaluated the influence of possible predictors on the BOP changes among all follow-up sessions.

DETAILED DESCRIPTION:
Fifty-six patients with 85 Implants affected by PM were randomly assigned to test (NSMD+FMD) or control procedures (NSMD + placebo). At baseline, 1, 3, 6 months, full-mouth plaque score (FMPS), full-mouth bleeding score (FMBS), probing depth (PD), bleeding on probing (BOP), modified gingival index (mGI), and modified plaque index (mPlI) were assessed. Furthermore, the proportions of Aggregatibacter Actynomycencomitans, Porphyromonas Gingivalis, Tannerella Forsythia and Treponema Denticola were also recorded. The BOP reduction was set as a primary outcome and the patient was considered statistical unit. Data were analysed to assess BOP reduction at a 6-month follow-up and to identify significant predictors of implant-site BOP through mixed generalized linear regression.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old;
* implants with smooth necks supporting cemented or screw-retained single-unit crowns with at least one BOP-positive site (Berglundh et al., 2018),
* implants placed in both maxilla and mandible
* patients with gingivitis or treated periodontitis with the absence of residual PD ≥5 mm
* presence at least of 2 mm of keratinized mucosa (KT) at implant sites

Exclusion Criteria:

* presence of systemic diseases;
* pregnancy or lactating;
* use of inflammatory drugs or antibiotics within 3 months prior to study recruitment;
* implants with modified (i.e., micro-rough) necks;
* interproximal open contacts between implant restoration and adjacent teeth;
* peri-implantitis (Berglundh et al., 2018)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) changes | 6-months
  The number of implants presenting with complete absence of BOP or implants with limited extent of BOP (≤1 spot/implant-the presence of a single spot)

SECONDARY OUTCOMES:
Probing pocket depth (PPD) changes | 6-months
  Changes in PPD
Full mouth plaque score (FMPS) % changes | 6-months
  Changes in FMPS%
Full mouth bleeding score (FMBS) % changes | 6-months
  Changes in FMBS%
Plaque at implant sites according to modified gingival index (mGI) changes score | 6-months
  Changes in mGI 0-4 score
Plaque at implant sites according to modified plaque index (mPlI) changes score | 6-months
  Changes in mPlI 0-4 score

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Results and clinical protocol
Supporting Information: Study Protocol
Time Frame: 6-months
Access Criteria: Official university website/pubmed